CLINICAL TRIAL: NCT01020942
Title: Cardioprotective of Electroacupuncture Pretreatment in Patients Underwent Coronary Stenting: A Prospective, Multicenter, Randomized Control Trial
Brief Title: Cardioprotective Effects of Electroacupuncture Pretreatment Against Coronary Stenting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XJMZK016
Record Dates: First submitted 2009-11-24; First posted 2009-11-26 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-11

CONDITIONS: Myocardial Injury
Keywords: ischemia; myocardial infarction; prognosis; pretreatment; electroacupuncture; stents; troponin; percutaneous coronary intervention
MeSH Terms: conditions — Ischemia; Myocardial Infarction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pretreatment (Experimental)
  Interventions: Procedure: Electroacupuncture stimulation
- Control (No Intervention)
  Interventions: Procedure: No intervention

INTERVENTIONS:
Procedure: Electroacupuncture stimulation — According to the theory of traditional Chinese medicine, bilateral Neiguan (PC 6) acupoints were chosen and identified according to traditional anatomical localizations. Once insertion of original needles was made at the acupoints, the needle was stimulated electrically with the intensity of 2-6 mA and frequency of 2/30 Hz using the Electronic Acupuncture Treatment Instrument until the patient felt the so-called 'Teh Chi' sensation of heaviness, numbness and swelling. The pretreatment was individualized based on patients sex, age, weight and felt and given 1 time per day for 5 consecutive days before the heart valve replacement surgery．
  Other Names: Preconditioning
  Arms: Pretreatment
Procedure: No intervention — The control patients were only placed needles at the bilateral Neiguan (PC 6)acupoints without electric stimulus.
  Other Names: Sham pretreatment
  Arms: Control

SUMMARY:
Myocyte necrosis as a result of elective percutaneous coronary intervention (PCI) occurs in approximately one third of cases and is associated with subsequent cardiovascular events. This study assesses the ability of electroacupuncture (EA) pretreatment to attenuate cardiac troponin I (cTnI) release after elective PCI.

DETAILED DESCRIPTION:
Elective percutaneous coronary intervention (PCI) is associated with troponin release in approximately one third of cases.Troponin release is a sensitive and specific marker of myocyte necrosis and infarction resulting from a form of ischemia/reperfusion injury, downstream embolization of atheromatous material, and coronary side-branch occlusion. A number of studies have demonstrated that procedure-related troponin release is associated with subsequent cardiovascular events.

Transient sublethal episodes of ischemia before a prolonged ischemia/reperfusion injury, known as ischemic preconditioning (IPC), have been shown to reduce the extent of myocardial infarction (MI).Electroacupuncture (EA) stimulus, as a pretreatment method, limits MI size in animal models. However, there are limited outcome to demonstrate protection from EA pretreatment during PCI. The present study investigated the ability of EA pretreatment to attenuate cardiac troponin I (cTnI) release after elective PCI in a single-center, randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* All patients > 18 of age who are undergoing elective PCI and are able to give informed consent are eligible for study.

Exclusion Criteria:

* Emergency PCI,
* Elevation of cTnI before PCI taken at the preadmission clinic,
* Women of child-bearing age,
* Nicorandil or glibenclamide use (preconditioning-mimetic and preconditioning blocking medication, respectively), and
* Severe comorbidity (estimated life expectancy < 6 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-12 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
The primary outcome was assessing whether EA pretreatment before elective PCI reduced cTnI concentration at 48 hours. | 48 hours after PCI

SECONDARY OUTCOMES:
Secondary outcomes were the effect of EA pretreatment on ischemic symptoms, ECG evidence of ischemia during coronary balloon occlusion, CRP,and major adverse cardiac events (MACE) at 6 months. | six months of PCI follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Lize Xiong, M.D., Ph.D., Study Director — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Wang Q, Liang D, Wang F, Li W, Han Y, Zhang W, Xie Y, Xin W, Zhou B, Sun D, Cao F, Xiong L. Efficacy of electroacupuncture pretreatment for myocardial injury in patients undergoing percutaneous coronary intervention: A randomized clinical trial with a 2-year follow-up. Int J Cardiol. 2015 Sep 1;194:28-35. doi: 10.1016/j.ijcard.2015.05.043. Epub 2015 May 13. PMID 26011261